CLINICAL TRIAL: NCT06493253
Title: Epidemiologic Liver Outcomes Retrospective Study to Confirm The Prognostic Value of the FibroNest Digital Pathology Fibrosis Biomarker (Ph-FCS) in Patients With MASLD (DPAILO-2)
Brief Title: Digital Pathology and AI for Liver Outcomes in MASLD (DPAILO-2)
Status: Not yet recruiting | Type: Observational
Sponsor: PharmaNest, Inc (Industry)
Collaborators: Nonalcoholic Steatohepatitis Clinical Research Network (NASH) (Unknown); Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Other Study IDs: PHN 1-020-24
Record Dates: First submitted 2024-07-02; First posted 2024-07-09 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Metabolic Dysfunction-associated Steatotic Liver Disease
Keywords: MASH

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Non-Liver Related Event: Absence of any of the liver events described in the second group in the patient clinical follow-up.
  Interventions: Diagnostic Test: Digital Pathology FibroNest Phenotypic Fibrosis Composite Score (Ph-FCS)
- Liver Related Event: Liver-related events include liver-related death, hepatic decompensation events (variceal hemorrhage, ascites, hepatic encephalopathy), and hepatocellular carcinoma.
  Interventions: Diagnostic Test: Digital Pathology FibroNest Phenotypic Fibrosis Composite Score (Ph-FCS)

INTERVENTIONS:
Diagnostic Test: Digital Pathology FibroNest Phenotypic Fibrosis Composite Score (Ph-FCS) — Biomarker name: FibroNest Phenotypic Fibrosis Composite Score Acronym: FibroNest Ph- FCS Type of Biomarker: Histologic based, Digital, Quantitative Image Analysis, Imaging modality Definition: A quantitative, normalized (no unit) and continuous composite

SUMMARY:
The aim of this multi-center, retrospective epidemiologic study is to confirm the prognostic performance of the Digital Pathology (DP) FibroNest Phenotypic Fibrosis Composite Score (Ph-FCS), derived from standard digital pathology liver biopsy images, in predicting clinical hepatic decompensation events in patients with metabolic dysfunction-associated steatohepatitis (MASH).

DETAILED DESCRIPTION:
MASH (Metabolic Dysfunction-Associated Steatohepatitis):

MASH presents histological liver changes similar to those caused by alcohol abuse, but occurs in the absence of alcohol intake. It is common among adults with conditions such as obesity and type-2 diabetes. Severe MASH is expected to become a leading cause of end-stage liver disease.

Current Challenges:

There are currently no fully approved treatments for MASH which places a significant burden on liver health and transplantation. Diagnosis and assessment rely on subjective histological reviews, which are prone to variability and limitations in detecting subtle changes. Therefore, there is an urgent need for accurate and continuous histological biomarkers.

FibroNest Ph-FCS Solution:

The FibroNest Ph-FCS offers a promising solution by utilizing high-resolution digital pathology and sophisticated algorithmic methods for sensitive and reproducible fibrosis severity assessment and prediction of clinical events. In a 2003 proof-of-concept retrospective study on 400 patients, the Ph-FCS demonstrated excellent prognostic performance.

Proposed Study:

This multi-center retrospective study aims to confirm the Ph-FCS's prognostic value using patient liver biopsies and clinical outcome data from the NAFLD Adult Database 2 registry (NCT01030484). The prognostic performance of the Ph-FCS will be compared to:

1. The NASH-CRN Histological Fibrosis Stages established from the same biopsies.
2. Non-invasive biomarkers like Fib-4 and elastography/Fibroscan, also collected retrospectively from the point of initial diagnosis.

Study Objectives:

(i) Confirm the Ph-FCS's prognostic utility on a large scale. (ii) Compare the Ph-FCS's prognostic performance with that of the NASH-CRN Fibrosis Stages established from the same biopsies.

(iii) Compare biopsy-based Ph-FCS with non-invasive biomarkers.

ELIGIBILITY:
From NCT01030484:

* Age at least 18 years during the consent process
* Willingness to be in the study for 1 or more years
* Ability and willingness to give written, informed consent to be screened for and, if eligible, to be enrolled into the Database 2 study
* Minimal or no alcohol use history consistent with NAFLD (see exclusion criteria)
* Collection of a liver biopsy that is obtained within 120 days of enrollment as part of standard of care or for evaluation in FLINT trial
* Collection of biosamples (serum, plasma, DNA, and, if available, liver tissue) within 90 days prior to enrollment and 0-90 days before or 4-90 days after the standard of care liver biopsy

Exclusion Criteria:

From NCT01030484

* Clinical or histological evidence of alcoholic liver disease or alcohol consumption during the two years before entry (> 20g/day for men, >10g/day women)
* History of total parenteral nutrition
* History of gastric or jejunoileal bypass preceding the diagnosis of NAFLD
* Biliopancreatic diversion or bariatric surgery
* Evidence of advanced liver disease with Child-Pugh-Turcotte score equal to or greater than 10
* Short bowel syndrome
* Suspected or confirmed hepatocellular carcinoma
* Positive for HIV
* Evidence of HBV or HCV infection
* Low alpha-1-antitrypsin level and ZZ phenotype
* Wilson's disease
* Known glycogen storage disease, dysbetalipoproteinemia, phenotypic hemochromatosis
* Vascular lesions
* Iron overload greater than 3+
* Zones of confluent necrosis, infarction, massive or sub-massive, pan-acinar necrosis
* Multiple epithelioid granulomas
* Congenital hepatic fibrosis
* Polycystic liver disease
* Other metabolic or congenital liver disease

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient from the NAFLD Adult Database 2 Registry including Adult pts ( >=18 years old) with MASLD defined histologically with >1 year of clinical follow up and available recording liver-related outcomes through clinical observation.
Sampling Method: Non-Probability Sample
Enrollment: 1700 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Performance of Hepatic Decompensation Event predictive value of the FibroNest Ph-FCS | Time-to-event analysis between 2 and 10 years
  Area under Receiver Operating Characteristic Curve (AUROC) of the FibroNest PT-Ph-FCS, as a prognostic/diagnostic biomarker for liver related events in patients with MASH.

SECONDARY OUTCOMES:
Performance of Hepatic Decompensation Event predictive value of the NASH-CRN Fibrosis Stage | Time-to-event analysis between 2 and 10 years
  Area under Receiver Operating Characteristic Curve (AUROC) of the NASH-CRN Fibrosis Stage, as a prognostic/diagnostic biomarker for liver related events in patients with MASH.
Performance of Hepatic Decompensation Event predictive value of the elastography (Fibroscan) biomarker, a non-invasive test | Time-to-event analysis between 2 and 10 years
  Area under Receiver Operating Characteristic Curve (AUROC) of the elastography (Fibroscan) biomarker, as a prognostic/diagnostic biomarker for liver related events in patients with MASH.

CONTACTS AND LOCATIONS:
Overall Officials: Arun J Sanyal, MD, Principal Investigator — Virginia Commonwealth University; Cynthia Belhling, MD, Study Director — University California San Diego; David E Kleiner, MD. PhD, Study Director — Nonalcoholic Steatohepatitis Clinical Research Network
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sanyal AJ, Van Natta ML, Clark J, Neuschwander-Tetri BA, Diehl A, Dasarathy S, Loomba R, Chalasani N, Kowdley K, Hameed B, Wilson LA, Yates KP, Belt P, Lazo M, Kleiner DE, Behling C, Tonascia J; NASH Clinical Research Network (CRN). Prospective Study of Outcomes in Adults with Nonalcoholic Fatty Liver Disease. N Engl J Med. 2021 Oct 21;385(17):1559-1569. doi: 10.1056/NEJMoa2029349. PMID 34670043
- [Background] Ratziu V, Chen L, Petitjean L. et al. Novel Artificial Intelligence-Assisted Digital Pathology Quantitative Image Analysis Predicts the occurrence of Liver-related Clinical Events in the Multicentric, European, Hepatic Outcomes and Survival Fatty Liver Registry (HITSURFR) Study. Hepatology. 78(S1) S1-S2154 2084-A
- Available data/document: Clinical Study Report: NCT01030484 — https://repository.niddk.nih.gov/studies/nafld-adult-database-2/ — The NAFLD Adult Database 2 continued the longitudinal follow-up of participants enrolled in earlier NASH CRN studies and recruited new participants with recent liver biopsies. Comprehensive data, including demographics, medical history, symptoms, medication use, alcohol use and routine laboratory studies were collected on all participants at entry and at annual visits for up to 10 years after enrollment. A liver biopsy was collected at baseline if not collected in a prior NASH CRN study.